CLINICAL TRIAL: NCT00034528
Title: Allogeneic Stem Cell Transplantation Following Nonmyeloablative Chemotherapy in Patients With Hemoglobinopathies
Brief Title: Stem Cell Transplantation After Reduced-Dose Chemotherapy for Patients With Sickle Cell Disease or Thalassemia
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Due to slow recruitment
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DAIT DF/HCC 01-098; P01 A 129530
Record Dates: First submitted 2002-04-30; First posted 2002-05-01 (Estimated); Last update posted 2013-05-01 (Estimated); Status verified 2013-04

CONDITIONS: Hemoglobinopathies; Anemia, Sickle Cell; Hemoglobin SC Disease; Thalassemia; Thalassemia Major
MeSH Terms: conditions — Hemoglobinopathies; Anemia, Sickle Cell; Hemoglobin SC Disease; Thalassemia; beta-Thalassemia | interventions — Busulfan; fludarabine; fludarabine phosphate; Tacrolimus; Prednisone

ARMS (1):
- Allogeneic stem cell transplantation (Experimental): Participants will receive a nonmyeloablative conditioning regimen of fludarabine and busulfan prior to allogeneic peripheral blood stem cell (CD34+) infusions. FK506 and prednisone will be administered for graft versus host disease (GVHD) prophylaxis.
  Interventions: Drug: Busulfan; Drug: Fludarabine; Drug: FK506; Drug: Prednisone

INTERVENTIONS:
Drug: Busulfan — 0.8 mg/kg/d administered as a single intravenous infusion over 3 hours for 4 days. All infusions are anticipated to be given in the outpatient clinic.
  Other Names: Busulfex
Drug: Fludarabine — 30 mg/m^2/d administered as a bolus infusion over 30 minutes for 4 days. All infusions are anticipated to be given in the outpatient clinic.
  Other Names: Fludara; Oforta
Drug: FK506 — 0.15 mg/kg taken orally daily for 12 to 14 weeks
  Other Names: Prograf; Tacromilus
Drug: Prednisone — 0.5 mg/kg taken orally four times daily on Day 7 and increase to 1 mg/kg taken orally four times daily on Day 14. Participants will continue regimen until Day 30 before a 20-25% taper per week.

SUMMARY:
The purpose of this study is to find out if using a lower dose of chemotherapy before stem cell transplantation can cure patients of sickle cell anemia or thalassemia while causing fewer severe side effects than conventional high dose chemotherapy with transplantation.

DETAILED DESCRIPTION:
Hemoglobinopathies, such as sickle cell disease and thalassemia major, are genetic diseases associated with significant morbidity and premature death. Allogeneic bone marrow transplantation (BMT) is the only potential cure for severe hemoglobinopathies. Typical regimens have used high doses of chemotherapy or chemo-radiotherapy to ablate recipient hematopoiesis and to prevent graft rejection. The widespread use of this treatment has been limited by toxicity, risk of end-organ damage, and donor availability. This study will use a nonmyeloablative regimen of fludarabine and busulfan to attempt to generate consistent engraftment with donor hematopoietic stem cells in patients with severe hemoglobinopathy.

G-CSF mobilization of the donor's peripheral blood white blood cells will precede donor apheresis. A nonmyeloablative conditioning regimen of fludarabine and busulfan will be administered to patients prior to allogeneic peripheral blood stem cell infusions. FK506 and prednisone will be administered for graft versus host disease (GVHD) prophylaxis. Patients will be evaluated for engraftment, donor: host hematopoietic chimerism, toxicity, and hemoglobinopathy.

ELIGIBILITY:
Inclusion criteria:

* All patients must:

  * Have related donors who are identical at 6 human leukocyte antigens (HLA) loci (A, B and DR) by molecular typing
  * Have a performance status from 0-2
  * Give written informed consent
* Patients with sickle cell disease should have 1 or more of the following:

  * Acute chest syndrome requiring recurrent hospitalization or exchange transfusion
  * Nonhemorrhagic stroke or central nervous system event lasting longer than 24 hours
  * Recurrent vaso-occlusive pain (2 episodes or more per year) or recurrent priapism
  * Sickle nephropathy (moderate or severe proteinuria or a glomerular filtration rate 30-50 percent of normal predicted value)
  * Bilateral proliferative retinopathy and major visual impairment in at least 1 eye
  * Osteonecrosis of multiple joints
* Patients with thalassemia should have 1 or more of the following:

  * Transfusion dependence, defined as a transfusion requirement of greater than or equal to 6 units of packed red blood cells over the past 12 months
  * Iron overload, defined as serum ferritin greater than 500 mcg/L in the absence of infection or biopsy-proven iron overload
  * Presence of 2 or more alloantibodies against red cell antigens

Exclusion criteria:

* Pregnancy
* Acute hepatitis (transaminases greater than 3 times the normal value)
* Cardiac ejection fraction less than 30 percent
* Severe renal impairment (glomerular filtration rate less than 30 percent of predicted normal value)
* Severe residual functional neurologic impairment (other than hemiplegia alone)
* Seropositivity for the human immunodeficiency virus (HIV)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2001-09; Primary Completion 2003-11 (Actual); Study Completion 2003-11 (Actual)

PRIMARY OUTCOMES:
Evidence of engraftment of donor hematopoietic cells following administration of low doses of busulfan and fludarabine | Throughout study

SECONDARY OUTCOMES:
Solid organ toxicity related to the conditioning regimen | Throughout study
Incidence of grade II, III, or IV acute graft versus host disease (GVHD) | Throughout study
Level of disease response | Throughout study

CONTACTS AND LOCATIONS:
Overall Officials: Catherine J. Wu, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (1):
- Dana-Farber Cancer Institute/Harvard Cancer Center, Brigham and Women's Hospital and Massachusetts General Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Background] Walters MC, Storb R, Patience M, Leisenring W, Taylor T, Sanders JE, Buchanan GE, Rogers ZR, Dinndorf P, Davies SC, Roberts IA, Dickerhoff R, Yeager AM, Hsu L, Kurtzberg J, Ohene-Frempong K, Bunin N, Bernaudin F, Wong WY, Scott JP, Margolis D, Vichinsky E, Wall DA, Wayne AS, Pegelow C, Redding-Lallinger R, Wiley J, Klemperer M, Mentzer WC, Smith FO, Sullivan KM. Impact of bone marrow transplantation for symptomatic sickle cell disease: an interim report. Multicenter investigation of bone marrow transplantation for sickle cell disease. Blood. 2000 Mar 15;95(6):1918-24. PMID 10706855
- [Background] Gomez-Almaguer D, Ruiz-Arguelles GJ, Ruiz-Arguelles A, Gonzalez-Llano O, Cantu OE, Hernandez NE. Hematopoietic stem cell allografts using a non-myeloablative conditioning regimen can be safely performed on an outpatient basis: report of four cases. Bone Marrow Transplant. 2000 Jan;25(2):131-3. doi: 10.1038/sj.bmt.1702100. PMID 10673669
- [Background] Krishnamurti L, Blazar BR, Wagner JE. Bone marrow transplantation without myeloablation for sickle cell disease. N Engl J Med. 2001 Jan 4;344(1):68. doi: 10.1056/NEJM200101043440119. No abstract available. PMID 11187121
- [Background] Andersson BS, Madden T, Tran HT, Hu WW, Blume KG, Chow DS, Champlin RE, Vaughan WP. Acute safety and pharmacokinetics of intravenous busulfan when used with oral busulfan and cyclophosphamide as pretransplantation conditioning therapy: a phase I study. Biol Blood Marrow Transplant. 2000;6(5A):548-54. doi: 10.1016/s1083-8791(00)70064-4. PMID 11071260
- [Background] Wu CJ, Krishnamurti L, Kutok JL, Biernacki M, Rogers S, Zhang W, Antin JH, Ritz J. Evidence for ineffective erythropoiesis in severe sickle cell disease. Blood. 2005 Nov 15;106(10):3639-45. doi: 10.1182/blood-2005-04-1376. Epub 2005 Aug 9. PMID 16091448
- [Background] Wu CJ, Gladwin M, Tisdale J, Hsieh M, Law T, Biernacki M, Rogers S, Wang X, Walters M, Zahrieh D, Antin JH, Ritz J, Krishnamurti L. Mixed haematopoietic chimerism for sickle cell disease prevents intravascular haemolysis. Br J Haematol. 2007 Nov;139(3):504-7. doi: 10.1111/j.1365-2141.2007.06803.x. No abstract available. PMID 17910640
- [Result] Wu CJ, Hochberg EP, Rogers SA, Kutok JL, Biernacki M, Nascimento AF, Marks P, Bridges K, Ritz J. Molecular assessment of erythroid lineage chimerism following nonmyeloablative allogeneic stem cell transplantation. Exp Hematol. 2003 Oct;31(10):924-33. doi: 10.1016/s0301-472x(03)00227-3. PMID 14550808